CLINICAL TRIAL: NCT04594187
Title: The Role of Nodal Radiation Therapy in Sentinel Lymph Node Positive Melanoma
Brief Title: Nodal Radiation Therapy for Sentinel Lymph Node Positive Melanoma
Acronym: MelPORT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0148; NCI-2020-06904 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0148 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-10; First posted 2020-10-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Immunotherapy; Adjuvants, Immunologic; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (immunotherapy, radiation therapy) (Experimental): Within 12 weeks of SLNB, patients start nodal radiation therapy (30 Gy in 5 treatments over 2-2.5 weeks). Immunotherapy planned to begin at any time after SLNB.
  Interventions: Other: Immunotherapy; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy
- Group II (immunotherapy) (Active Comparator): Patients planned to undergo immunotherapy.
  Interventions: Other: Immunotherapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Immunotherapy — All patients must be planned for treatment with any immunotherapy agent after sentinel lymph node biopsy (e.g. pembrolizumab or nivolumab). For patients receiving radiation therapy initiation may be before, during or after radiation.
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo nodal radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group I (immunotherapy, radiation therapy)

SUMMARY:
This phase II trial seeks to determine the role of nodal radiation therapy after sentinel lymph node biopsy (SLNB) for patients with high risk sentinel lymph node positive melanoma who are planned for immunotherapy without completion lymph node dissection. Prior studies of patients with more advanced melanoma have shown nodal radiation therapy can decrease the risk of nodal recurrence but it is not known if this same benefit will be seen in patients with high risk sentinel lymph node positive disease who are planned for immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if regional nodal radiation therapy prolongs the time to regional recurrence.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive adjuvant immunotherapy and nodal radiation therapy (30 Gy in 5 treatments over 2-2.5 weeks).

GROUP II: Patients receive adjuvant immunotherapy alone.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be planned for post-operative immunotherapy
* No evidence of distant metastasis as determined by clinical examination and any form of imaging
* No evidence of clinically involved lymph nodes prior to SLNB
* Pathologically confirmed sentinel lymph node positive melanoma with high risk features (extracapsular extension [ECE] or 0.5 mm+ nodal tumor implant or 2+ involved nodes or lymphovascular invasion of the primary tumor)
* Has provided written informed consent for participation in this trial
* Eastern Cooperative Oncology Group (ECOG) performance status of 3 or less
* Life expectancy greater than 6 months
* Patients capable of childbearing are using adequate contraception
* Available for follow-up

Exclusion Criteria:

* Complete lymph node dissection (CLND) of the nodal basin containing the positive SLN
* Distant metastasis
* Previous radiation therapy (RT) to the nodal area planned for RT such that the prior RT field would be included in the current treatment field. In other words, treatment on this trial would require re-irradiation of tissues
* Women who are pregnant
* Adults unable to consent, individuals who are not yet adults, pregnant women and prisoners will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to regional nodal recurrence | From date of sentinel lymph node biopsy, assessed up to 5 years
  Regional nodal recurrence will be assessed by physical exam and routine surveillance imaging during follow-up

SECONDARY OUTCOMES:
Time to locoregional recurrence | From date of sentinel lymph node biopsy, assessed up to 5 years
  Local recurrence, locoregional recurrence (including both regional recurrence and local recurrence at the primary tumor site) will also be assessed by physical exam and routine surveillance imaging during follow-up.
Time to distant metastasis | From date of sentinel lymph node biopsy, assessed up to 5 years
  Distant metastasis will also be assessed by physical exam and routine surveillance imaging during follow-up.
Progression-free survival | From date of sentinel lymph node biopsy to recurrence event or last follow-up, assessed up to 5 years
Overall survival | From date of sentinel lymph node biopsy to last follow-up, assessed up to 5 years
Incidence of long term toxicity | Up to 5 years
  Long term toxicity including lymphedema, infection, decreased mobility will be assessed at the time of routine follow up appointments. Physician-reported toxicity related to regional nodal disease or treatment will be recorded as per Common Terminology Criteria for Adverse Events version 5.0. Specific toxicity to be evaluated will include: fatigue, localized edema, lymphedema, pain, skin infection, soft tissue infection, thrush, radiation recall reaction, arthritis, fibrosis, joint range of motion, dysphagia, dysgeusia and dry skin.
Patient reported quality of life | At baseline, 3 months after sentinel lymph node biopsy, 9 months after sentinel lymph node biopsy, and 2 years after sentinel lymph node biopsy
  Quality of life in all patients will be assessed by Functional Assessment of Cancer Therapy General survey. Patients with head and neck nodal disease will also be assessed by the University of Washington Quality of Life survey and patients with axillary nodal disease will also be assessed by the Lymphoedema Quality of Life-ARM.

OTHER OUTCOMES:
Tissue associated biomarkers of disease control and radiation-associated toxicity | Up to 5 years
Optional blood associated biomarkers of disease control and radiation-associated toxicity | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Devarati Mitra, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Cooper Hospital UNIV MED CTR., Camden, New Jersey
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org